CLINICAL TRIAL: NCT00001253
Title: Estrogen Effects on Cognition in Girls With Turner Syndrome
Brief Title: The Effects of Estrogen on Cognition in Girls With Turner Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 900123; 90-CH-0123
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-03

CONDITIONS: Gonadal Dysgenesis; Turner's Syndrome
Keywords: Turner's Syndrome; Estrogen; Ethinyl estradiol; Learning; Ovarian dysgenesis
MeSH Terms: conditions — Gonadal Dysgenesis; Turner Syndrome | interventions — Neuropsychological Tests; Weights and Measures

INTERVENTIONS:
Behavioral: cognitive tests and scales

SUMMARY:
The development of the brain in females is a result of a combination of factors. During puberty estrogen plays a role in influencing brain development. Cultural and environmental factors also play a role in the development of the brain.

Female patients with Turner syndrome lack the ability to produce estrogen due to undeveloped ovaries. Therefore, Turner syndrome is the perfect condition to study how estrogen (or the lack of estrogen) influences a person's behavior and thinking.

This study will compare cognitive differences (visual motor skills, visual-spatial, psychosocial behavior, and visual memory) of patients with Turner syndrome to normal patient controls. Researchers will use the Weschler Intelligence Scale for Children-Revised (WISC-R) along with other tests and scales to measure different aspects of the patient's cognitive ability. In addition the study will review patients with Turner syndrome who previously received estrogen replacement as infants and children in a related research study.

Researchers hope to demonstrate that estrogen replacement will improve cognition and behavior in girls with Turner syndrome.

DETAILED DESCRIPTION:
Estrogen influences brain development in females at puberty. Environmental and cultural factors interact with the biological effects of estrogen on the brain and consequently on cognition and behavior. Turner syndrome females lack endogenous estrogen as a result of dysgenetic ovaries. Turner syndrome therefore represents a unique, estrogen-deficient model in which to study the biological effects of estrogen on cognition and behavior. The specific aims of this project are to: 1) document further, the cognitive differences between girls with Turner syndrome at ages 5 to adult (less than or equal to age 50) versus age-matched, female controls. 2) to examine the differential effects of continuous estrogen replacement in infancy and in early childhood on cognitive and social function in a unique, previously approved, randomized, double-blind, placebo-controlled, treatment trial (87-CH-0152). Specifically, we hypothesize that estrogen replacement in early childhood will reduce the cognitive deficits of girls with Turner syndrome. In addition, we hypothesize that the degree of socialization ability in these girls will correlate with social-behavioral and social recognition ability. Finally, we hypothesize that earlier (infancy to 8 years) and longer estrogen replacement will result in less impairment of visual-motor ability, visual-spatial ability, socialization ability, and affective competence compared to later (9 to 12 years) estrogen replacement in girls with Turner syndrome.

Children with Turner syndrome and controls will be tested in the Outpatient Departments at the two approved sites of protocol 87-CH-0152; the NIH and Thomas Jefferson University.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients will include girls and women ages 5-50 yr with the diagnosis of Turner syndrome based on absence of all or part of one of the X chromosomes.

Control subjects must be within +/- 2SD for height and weight and have normal intelligence and educational achievement.

Biological parents (both male and female) of TS subjects may be included in this study, but only to have blood drawn for genetic testing in order to determine the origin of the X-chromosome of their daughters.

EXCLUSION CRITERIA:

Those with severe physical or neurocognitive impairment, preventing accurate completion of the cognitive tasks, will be excluded.

Normal subjects who have qualified for or participated in gifted and talented or remedial education programs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 950
Dates: Start 1990-05; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Palmer CG, Reichmann A. Chromosomal and clinical findings in 110 females with Turner syndrome. Hum Genet. 1976 Dec 29;35(1):35-49. doi: 10.1007/BF00295617. PMID 1002163
- [Background] Singh RP, Carr DH. The anatomy and histology of XO human embryos and fetuses. Anat Rec. 1966 Jul;155(3):369-83. doi: 10.1002/ar.1091550309. No abstract available. PMID 5956901
- [Background] Park E, Bailey JD, Cowell CA. Growth and maturation of patients with Turner's syndrome. Pediatr Res. 1983 Jan;17(1):1-7. doi: 10.1203/00006450-198301000-00001. No abstract available. PMID 6835711